CLINICAL TRIAL: NCT05461456
Title: An Open Label, Single-Dose, Single-Treatment, Single-Period Safety and Bioavailability Study of Fexofenadine Hydrochloride Topical Lotion 1% in Healthy, Adult, Male Human Subjects
Brief Title: Bioavailability and Tolerability of Fexofenadine Hydrochloride Topical Lotion 1%
Acronym: ATOFEX-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OrchestratePharma GmbH (Industry)
Collaborators: VidiLife Clinical Research Associate (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iVRS-CD-22-021
Record Dates: First submitted 2022-07-02; First posted 2022-07-18 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis Eczema; Atopic Rash; Rash; Pruritus; Urticaria; Urticaria Chronic; Psoriasis; Psoriasis Vulgaris; Skin Rash; Skin Inflammation; Eczema
Keywords: Inflammatory Skin Disease; Pruritus; Rash; Atopic Dermatitis; Urticaria; Psoriasis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Exanthema; Pruritus; Urticaria; Chronic Urticaria; Psoriasis; Dermatitis; Eczema

STUDY DESIGN:
Intervention Model Description: The study is an 'Open Label, Single-Dose, Single-Treatment, Single-Period Safety and Bioavailability Study in Healthy, Adult, Male Human Subjects, where the subjects will be housed in the clinical facility from not less than 11 hours pre-dose till at least 72 hours post-dose. Altogether, the subject will stay for consecutive 03 days and 04 nights in the facility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OP2101 (Experimental): Treatment with Fexofenadine Hydrochloride Topical Lotion 1% (OP2101)
  Interventions: Drug: Fexofenadine Hydrochloride Topical Lotion 1% (OP2101)

INTERVENTIONS:
Drug: Fexofenadine Hydrochloride Topical Lotion 1% (OP2101) — Intervention:
  The amount of study lotion (OP2101) used is 11 grams per subject, equivalent to 22 fingertip units (FTU). The lotion is applied to the subject on back and front of the trunk, both hands (palm and back) and both arms. An SOP for handling and application of the lotion ensures the 11 grams covers 54% of the body surface area (BSA) evenly without residue.
  Comment:
  The treatment is single-dose and single-treatment. The FTU is used to standardize the amount of cream being applied in clinical research. It is also used in clinical practice and hence connects the objectiveness of the trial to the clinical situation.

SUMMARY:
The investigational lotion is envisaged as an short- and long term "Ease & Prevent" monotherapy for adults and children with mild to moderate eczema. With itch representing the most burdensome symptom in eczema, the main objectives with the lotion is fast and efficient itch relief, high tolerability, and high short- and long term safety. This phase 1 study aims to monitor skin tolerability, and how much of the active compound that is absorbed to the bloodstream.

DETAILED DESCRIPTION:
Fexofenadine Hydrochloride Topical Lotion 1% (OP2101) is a novel formulation developed for the treatment of skin disorders characterized by pruritus. Research show that oral Fexofenadine Hydrochloride (FX) may lead to a small improvement of pruritus in patients with Atopic Dermatitis (AD). In clinical practice, oral antihistamines are widely used off-label for pruritus relief in AD, indicating a discrepancy in trial outcomes and real-life experience. The pre-study thesis postulates that the antipruritic effect of FX can be leveraged in a dose-response relationship facilitated by high topical concentration of FX in direct contact with the pathological process of the skin. The sponsor also suggest that the Cytosolic phospholipase A2 (cPLA2) blocking property of FX is an untapped resource that is likely to be dose-response dependent and manifested by means of high topical concentration in proximity to the inflammatory process. The repositioning of FX to a topical treatment has the potential for high safety, efficacy, fast relief, and ease of use. OP2101 is also aimed at inflammation control, suppression of bacterial imbalance, moisture retention, upregulation of antimicrobial peptides, and skin barrier restoration. As such, it targets six of the pathological pillars of AD. Assessment of topical tolerability and skin adsorption (systemic exposure) are the main objectives in this phase 1 study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male human subjects between 18 to 45 years of age (both inclusive).
2. Having a Body Mass Index (BMI) between 18.5 and 30.0 kg/m2 (both inclusive).
3. Have no abnormal findings during screening done 21 days prior to administration of study drug, medical history and examination, laboratory evaluations, 12-lead ECG recordings.
4. Has an optimum physical condition which enables subjects to be fit for a Pharmacokinetic sampling according to principal investigator's evaluation.
5. Able to comply with the study procedures in the opinion of the PI/CI.
6. Able to give written consent for participation in the study.
7. Subjects who have taken at least two doses of COVID 19 vaccine and possess certificate for the same.
8. Intact skin without major scarring or tattoos.
9. An unusual diet (e.g., low salt), for any medical reason or non-medical reason for three weeks prior to receiving the study drug and throughout the subjects' participation in the study. In any such case subject selection will be at the discretion of the PI/CI.

Exclusion Criteria:

1. Known hypersensitivity or idiosyncratic reaction to Fexofenadine Hydrochloride or any of the excipients in the formulation.
2. Diagnosed with, or a family history of, long QT syndrome (LQTS).
3. Skin disorders or current skin discomforts.
4. Any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal, genital or any other body system.
5. Ingestion of any medicine at any time within 14 days before Check In. In any such case subject selection will be at the discretion of the PI/CI and medicine taken will be recorded.
6. Any history or presence of asthma (including aspirin induced asthma) or NSAID induced urticaria.
7. History of substance abuse and or addiction to drugs and alcohol.
8. Smokers, who smoke 9 or more cigarettes / day or inability to abstain during the study.
9. Habituated to drinking tea or coffee (more than 5 cups/day) or inability to abstain during the study
10. Habituated to tobacco/tobacco containing products (more than 10 gm/day) or inability to abstain during the study.
11. A positive result for Serological tests [including hepatitis B & C, HIV antibody and syphilis {VDRL (RPR) /TPHA}] tests.
12. Donation of blood (1 unit: 350 mL) within 90 days prior to receiving the first dose of study drug.
13. The receipt of an investigational product or participation in a drug research study within a period of 90 days prior to the first dose of study drug.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2022-10-16 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 0-72 hours
  Incidence and severity of local and systemic Adverse Events (AEs).
Cmax | 0.00 (pre-dose) and at 1.00, 4.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 60.00- & 72.00-hours post-dosing.
  Peak plasma concentration (Cmax)
Tmax | 0.00 (pre-dose) and at 1.00, 4.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 60.00- & 72.00-hours post-dosing.
  Peak plasma time (Tmax)
T½ | 0.00 (pre-dose) and at 1.00, 4.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 60.00- & 72.00-hours post-dosing.
  Half-life (T½)
AUC0-72h | 0.00 (pre-dose) and at 1.00, 4.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 60.00- & 72.00-hours post-dosing.
  Area under the curve (AUC0-72h)

SECONDARY OUTCOMES:
Dermal tolerability and treatment perception | -60 minutes, 30 minutes, 72 hours
  Skin- and Lotion Assessment Questionnaire (SLAQ) is a proprietary 3-part questionnaire:
  * Part 1 is a 6-modalities, 4-grade self-assessment of skin perceptions.
  * Part 2 is the Local Tolerability Scale (LTS).
  * Part 3 is a 7-modalities, 5-grade assessment of cream properties.

OTHER OUTCOMES:
Radial pulse | At the time of check-in, prior to dosing and at 03.00, 06.00, 12.00, 24.00, 36.00, 48.00, & 60.00 hours (± 60 minutes) post dose and prior to check-out.
  Radial pulse (beats per minute)
Systolic blood pressure | At the time of check-in, prior to dosing and at 03.00, 06.00, 12.00, 24.00, 36.00, 48.00, & 60.00 hours (± 60 minutes) post dose and prior to check-out.
  Systolic blood pressure (mmHg)
Diastolic blood pressure | At the time of check-in, prior to dosing and at 03.00, 06.00, 12.00, 24.00, 36.00, 48.00, & 60.00 hours (± 60 minutes) post dose and prior to check-out.
  Diastolic blood pressure (mmHg)
Respiratory rate | 0.00 (pre-dose) and at 1.00, 4.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 60.00- & 72.00-hours post-dosing.
  Respiratory rate (breaths per minute)
Body temperature | 0.00 (pre-dose) and at 1.00, 4.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 60.00- & 72.00-hours post-dosing.
  Body temperature (Celsius degrees)

CONTACTS AND LOCATIONS:
Locations (1):
- BCT Ltd., Dhaka, Ramna, Bangladesh